CLINICAL TRIAL: NCT06261229
Title: The Effectiveness of Intermittent Fasting and Behavioral Economics Intervention on Weight Control in Obese Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2022/230
Record Dates: First submitted 2022-10-04; First posted 2024-02-15 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Intermittent Fasting; Weight Loss; Behavioral Economic; Obese; HOMA-IR
Keywords: Intermittent Fasting; behavioral economic; Obese patients; Weight control; HOMA-IR
MeSH Terms: conditions — Intermittent Fasting; Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent fasting (Experimental): The participant will consume food about/ within 8 hours per day
  Interventions: Behavioral: Intermittent fasting
- Intermittent fasting + Behavioral economic (Experimental): The participant will consume food about/ within 8-hour per day. They will be rewarded as money when they achieve their weight loss goal or/and successfully do intermittent fasting 5 days/week.
  Interventions: Behavioral: Intermittent fasting + Behavioral economic
- Intensive Lifestyle Modification (Experimental): Advice about nutrition knowledge, healthy eating diet, diet prescription, and exercise
  Interventions: Behavioral: Intensive Lifestyle Modification

INTERVENTIONS:
Behavioral: Intermittent fasting — The participant will consume food about/ within 8-hour per day
  Arms: Intermittent fasting
Behavioral: Intermittent fasting + Behavioral economic — The participant will consume food about/ within 8-hour per day. They will be received a reward as money when achieve weight loss goal or/and success doing intermittent fasting 5 days/week
  Other Names: Intermittent fasting + Incentives
  Arms: Intermittent fasting + Behavioral economic
Behavioral: Intensive Lifestyle Modification — Advice about nutrition knowledge, healthy eating diet, diet prescription, and exercise
  Arms: Intensive Lifestyle Modification

SUMMARY:
This study is a parallel randomized controlled trial (RCT). To determine the effect of intermittent fasting, intermittent fasting with behavioral economics, and intensive lifestyle modification on nutritional status; the differences between HOMA-IR, body weight change, and body composition in obese people.

Each participant will be randomized to receive the intervention (intermittent fasting, intermittent fasting with behavioral economics, or intensive lifestyle modification.

The study protocol will be explained to the eligible participant and informed written consent will be obtained.

The total sample size will be 123 participants. Blood and urine samples will be collected at baseline and each follow-up visit including 1-month, 2-months, 6-month, and 12-months, respectively for further study to find out the mechanisms of weight loss, weight regain, and the improvement in the metabolic disease.

DETAILED DESCRIPTION:
The investigators will collect the participant characteristics (age, gender, smoking history, comorbid diseases including history of previous stroke, myocardial infarction, angina, hypertension, dyslipidemia, T2DM, risk of osteoporosis, and all medication lists) at the first visit.

* Physiological parameters:

  1. Body composition will be assessed by the Bioelectrical Impedance at the first visit and at each follow-up visit (1 month, 2 months, 4 months, 6 months, 9 months, and 12 months).
  2. Peripheral venous blood sample (15mL: clotted blood 9mL and EDTA blood 6 mL) and urinalysis will be collected from all participants at baseline and each follow-up visit (1-month, 2-months, 6-month, and 12 months). Blood samples will be immediately centrifuged and plasma/serum will be placed in a -80 Celsius freezer until analysis (glucose, HbA1C, insulin, albumin, creatinine, uric acid, lipid profile, liver function test, kidney function test, thyroid function test, and other biochemical).
* Three questionnaires will be collected:

  1) Global physical activity questionnaire, sleep questionnaire, and satiety visual analog score questionnaire will be obtained at the first visit and at each follow-up visit (1 month, 2 months, 4 months, 6 months, 9 months, and 12 months).
* Nutritional status will be assessed by history, 24-hour dietary recall, 3days food record, and physical examinations at the first visit and at each follow-up visit (1 month, 2 months, 4 months, 6 months, 9 months, and 12 months).

Regarding the descriptive statistical analysis, all the data will be tested for normality. Data will be presented as Mean ± standard deviation or Median (interquartile ranges) for continuous variables and frequency (%) for binary and categorical variables. The continuous variables will be compared by using Independent samples T-test or Analysis of variance (ANOVA) followed by multiple comparisons with the Bonferroni method. Test results of categorical variables will be evaluated by Chi-square or Fisher exact test as appropriate. Results will be deemed statistically significant at a P-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 year
* BMI start at 25.0 kg/m2 (above 24.99 kg/m2)
* Weight change less than 5% in 6-month
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Pregnant women or breed feeding
* Kidney disease/ Liver disease
* Abnormal Thyroid hormone, abnormal GI function
* Postoperative bariatric surgery
* Drug control weight or reduce appetite
* Drug abuse
* Mental illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
HOMR-IR (index) | Change from Baseline HOMR-IR at 6 months and 12 months
  Homeostatic Model Assessment for Insulin Resistance
Body mass index (kg/m^2) | Change from Baseline Body mass index at 1 month, 2 months, 4 months, 6 months, 9 months, and 12 months
  Body weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
FBS (mg/dl) | Change from Baseline FBS (mg/dl) at 1 month, 2 months, 6 months, and 12 months
  Fasting blood glucose
HbA1C (%) | Change from Baseline HbA1C (%) at 1 month, 2 months, 6 months, and 12 months
  Average blood sugar levels over the past 3 months
Albumin (g/L) | Change from Baseline Albumin (g/L) at 1 month, 2 months, 6 months, and 12 months
  a blood plasma protein synthesized in the liver
Creatinine (mg/dL) | Change from Baseline Creatinine (mg/dL) at 1 month, 2 months, 6 months, and 12 months
  a waste product that comes from the normal wear and tear on muscles of the body
Alanine transaminase (ALT) U/L | Change from Baseline Alanine transaminase (ALT) U/L at 1 month, 2 months, 6 months, and 12 months
  ALT is commonly measured clinically as part of liver function tests
Aspartate transaminase (AST) U/L | Change from Baseline Aspartate transaminase (AST) U/L at 1 month, 2 months, 6 months, and 12 months
  AST is commonly measured clinically as part of liver function tests
Uric acid (mg/dL) | Change from Baseline Uric acid (mg/dL) at 1 month, 2 months, 6 months, and 12 months
Total cholesterol (mg/dL) | Change from Baseline Total cholesterol (mg/dL) at 1 month, 2 months, 6 months, and 12 months
HDL-C (mg/dL) | Change from Baseline HDL-C (mg/dL) at 1 month, 2 months, 6 months, and 12 months
  High-density lipoprotein cholesterol
LDL-C (mg/dL) | Change from Baseline LDL-C (mg/dL) at 1 month, 2 months, 6 months, and 12 months
  Low-density lipoprotein cholesterol
Triglycerides (mg/dL) | Change from Baseline Triglycerides (mg/dL) at 1 month, 2 months, 6 months, and 12 months
Blood Urea Nitrogen (BUN) (mg/dL) | Change from Baseline Blood Urea Nitrogen (BUN) (mg/dL) at 1 month, 2 months, 6 months, and 12 months
Urine albumin-creatinine ratio (UACR) (mg/g) | Change from Baseline Urine albumin-creatinine ratio (UACR) (mg/g) at 1 month, 2 months, 6 months, and 12 months
Energy from food (kilocalories) | Change from Baseline Energy from food (kilocalories) at 1 month, 2 months, 4 months, 6 months, 9 months, and 12 months
  Energy from food (kilocalories) assess by 24hour-dietary recall and 3days food record

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No